CLINICAL TRIAL: NCT06687473
Title: The Study of Bismuth Salt Effect on the Virulence Factors of Helicobacter Pylori and Its Therapeutic Role for Multiple-resistant Strains
Brief Title: Susceptibility-guided Bismuth Quadruple Therapy for Multiple-resistant Helicobacter Pylori Strains
Acronym: BSUS-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-110-096
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Helicobacter Pylori; Drug Resistance, Multiple; Virulence Factor
Keywords: bismuth; microbial sensitivity tests; Helicobacter pylori; drug resistance, multiple; Virulence Factor

STUDY DESIGN:
Intervention Model Description: The multi-resistant H. pylori eradication rates between "bismuth-susceptibility-based regimen" and history "physicians' discretion regimen" are compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bismuth-based susceptibility-guided treatment (Experimental): Participants who have triple- or quadruple-drug resistant H. pylori infection are enrolled. Participants receive one of the four regimens based on susceptibility test.
  Interventions: Drug: Bismuth-based susceptibility-guided treatment

INTERVENTIONS:
Drug: Bismuth-based susceptibility-guided treatment — The investigators design four regimes for H. pylori eradication and participants receive one of the regimens based on susceptibility test. The four regimens are PBAT for those with both amoxicillin and tetracycline susceptible H. pylori; PBAM for those with amoxicillin susceptible but tetracycline resistant H. pylori; PBMT for those with amoxicillin resistant but tetracycline susceptible H. pylori; PBMR for those with both amoxicillin and tetracycline resistant H. pylori.
  A is amoxicillin (1000 mg thrice daily), B is colloidal bismuth subcitrate (120 mg thrice daily), M is metronidazole (500 mg thrice daily), P is a proton pump inhibitor, i.e., esomeprazole (40 mg twice daily), R is rifabutin (150 mg twice daily), and T is tetracycline (500 mg thrice daily). The treatment duration is 14 days for all regimens.

SUMMARY:
The goal of this clinical trial is to learn if the 14-day susceptibility-guided bismuth quadruple therapy works to treat multiple drug resistant Helicobacter pylori (H. pylori) in adults. It will also learn about the adverse effects of bismuth quadruple therapy. The main questions it aims to answer are:

* Does 14-day susceptibility-guided bismuth quadruple therapy higher the eradication rate?
* What medical problems do participants have when taking 14-day susceptibility-guided bismuth quadruple?
* Does bismuth suppress the expression of virulence factors of H. pylori?

Researchers will record 14-day susceptibility-guided bismuth quadruple to see if 14-day susceptibility-guided bismuth quadruple works to treat multiple drug resistant H. pylori.

Participants will:

* Take susceptibility-guided bismuth quadruple every day for 14 days
* Visit the clinic once 4-6 weeks for checkups and tests
* Keep a diary of their symptoms during taking susceptibility-guided bismuth quadruple

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infection is the major culprit of dyspeptic symptoms, peptic ulcer disease, gastric adenocarcinoma, and gastric mucosa-associated lymphoid tissue lymphoma. The Tokyo consensus stated that infection with H. pylori should be regarded as a pathogenic infectious disease rather than commensals only and should be eradicated.

H. pylori eradication regimen evolved with the increase of resistance rate in different regions. In Taiwan, clarithromycin resistance rate is arising from 9.5% in 2009 to around 14-17% in 2016 when conducting the first-line therapy. As a result, Taiwan gastroenterological association consensus suggested using 14-day clarithromycin-based (hybrid, sequential, concomitant, or triple) therapy as the first-line therapy and levofloxacin-based therapy as the second line therapy according to endemic resistance rate.

After twice eradication failure, H. pylori culture for susceptibility test is strongly recommended, which guide clinician to choose appropriate susceptibility-based therapy. Progressive increased dual (clarithromycin and levofloxacin) resistance and triple (dual and metronidazole) resistance, however, made it difficult for eradication. The regimens at physicians' discretion varied a lot and the overall successful eradication rate around 60% was still unsatisfactory.

Susceptibility-guided therapy is currently the consensus recommendation for 3rd-line H. pylori eradication. Bismuth quadruple therapy could overcome either clarithromycin or metronidazole resistant strains. Several evidences of clinical randomized-controlled trials demonstrated that adding bismuth as the first line therapeutic regimen can capture additional 30-40% successful eradication rate for the resistant strain, further contributing to the overall eradication rate. Accordingly, the aim of our study was to validate the susceptibility-guided bismuth quadruple therapy in patients with multiple drug resistant H. pylori infection in terms of efficacy and side effects.

Almost more than 99.5% ingested bismuth salt can be excreted from intestinal lumen without absorption. Bismuth may be able to form complexes in bacterial wall and periplasmic space, as well as inhibits enzymes, ATP synthesis and bacterial adherence to gastric mucosa. The MIC90 of bismuth to Helicobacter pylori ranged from 4-32 ng/L and there was no resistance been reported. Lots of H. pylori virulence factors are important players to establish colonization in gastric environment in each steps. Urease activity adjusts the pericellular environment to less acidity. Flagella direct bacterial motility and chemotaxis to mucosal surface. Colonization to epithelium is facilitated by lots of adhesion-receptor interaction, including BabA to Lewis B, SabA to sialyl-Lewis X, and CagL to α5β1 integrin. Bismuth drugs may affect the urease activity in jack bean plant and Klebsiella aerogenes. Bismuth inactivates H. pylori nickel-responsive transcription factor (NikR) protein, an important regulator for nickel homeostasis and iron metabolism in H. pylori. Since nickel iron is crucial in the catalytic function of urease, it is reasonable to assuming that it may impose effect on the urease activity in H. pylori. Furthermore, a pilot study showed that nickel-free diet can enhance the H. pylori eradication rate, which was speculated due to decreased urease activity.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori-infected with treatment experience with at least one course of eradication failure
* H. pylori-infected with treatment naïve but having multiple-drug resistant H. pylori (>= three antibiotics)
* H. pylori infection confirmed by H. pylori culture

Exclusion Criteria:

* Previous allergic reactions to regimens, including amoxicillin, bismuth subcitrate, esomeprazole, metronidazole, rifabutin, and tetracycline,
* Severe comorbidities,
* Chronic kidney disease with estimated glomerular filtration rate < 60 ml/min/1.73 m2,
* Pregnant or breastfeeding women.
* Dual-resistant H. pylori infection
* Mono-resistant H. pylori infection
* All susceptible H. pylori infection
* Positive RUT but negative H. pylori culture
* Negative RUT and negative H. pylori culture
* Decline to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The eradication rate of H. pylori | From enrollment to the end of treatment at 6-8 weeks
  The investigators define successful eradication as a negative 13C-urea breath test or a negative H. pylori stool antigen test at 4 to 6 weeks after the completion of H. pylori eradication and discontinuation of antibiotics and proton pump inhibitors. The eradication rates are determined by intention-to-treat and per-protocol analyses. The intention-to-treat analysis evaluates all enrolled participants. The per-protocol analysis evaluates those who take >= 80% of the study medications and receive post-treatment 13C-urea breath test or an H. pylori stool antigen test. The successful rate is represented with a percentage (%).

SECONDARY OUTCOMES:
Adverse effects | From enrollment to the end of treatment at 2 weeks
  Adverse events are assessed by a physician and a format questionnaire survey after the end of treatment. Serious adverse events are defined as daily activities restricted or participant unable to work. The adverse events include dizziness, skin rash, headache, unpleasant taste/bitter, abdominal pain, nausea, vomiting, diarrhea, constipation, abdominal fullness, glossitis/sore throat, darkened stool, fatigue, anorexia, chest burn, palpitation, and vaginal discharge. All adverse events are classified as none, mild (not restricting daily activities), or serious (restricting daily activities or causing inability to work).
Adherence to medications | From enrollment to the end of treatment at 2 weeks
  Adherence to medications is evaluated by questionnaire surveys after treatment completion. Adherence of medications is categorized as good (≥ 80% medication taken) or poor (< 80% medication taken).

OTHER OUTCOMES:
The sex-based eradication rate of H. pylori | From enrollment to the end of treatment at 6-8 weeks
  The eradication rates are evaluated in females and males, respectively. The investigators define successful eradication as a negative 13C-urea breath test at least four weeks after the completion of H. pylori eradication and discontinuation of antibiotics and proton pump inhibitors. The eradication rates are determined by ITT and PP analyses. The ITT analysis evaluates all enrolled participants. The PP analysis evaluates those who take >= 80% of the study medications and receive post-treatment 13C-urea breath test. The staffs assessing antibiotic sensitivity and the 13C-urea breath test are blinded.
The regimen-based eradication rate of H. pylori | From enrollment to the end of treatment at 6-8 weeks
  The eradication rates are evaluated in the four regimens, respectively. The investigators define successful eradication as a negative 13C-urea breath test at least four weeks after the completion of H. pylori eradication and discontinuation of antibiotics and proton pump inhibitors. The eradication rates are determined by ITT and PP analyses. The ITT analysis evaluates all enrolled participants. The PP analysis evaluates those who take >= 80% of the study medications and receive post-treatment 13C-urea breath test. The staffs assessing antibiotic sensitivity and the 13C-urea breath test are blinded.
The resistance-number-based eradication rate of H. pylori | From enrollment to the end of treatment at 6-8 weeks
  The eradication rates are evaluated in the subjects with triple-resistant infection and those with quadruple-resistant infection, respectively. The investigators define successful eradication as a negative 13C-urea breath test at least four weeks after the completion of H. pylori eradication and discontinuation of antibiotics and proton pump inhibitors. The eradication rates are determined by ITT and PP analyses. The ITT analysis evaluates all enrolled participants. The PP analysis evaluates those who take >= 80% of the study medications and receive post-treatment 13C-urea breath test. The staffs assessing antibiotic sensitivity and the 13C-urea breath test are blinded.
The treatment-failure-experience-based eradication rate of H. pylori | From enrollment to the end of treatment at 6-8 weeks
  The eradication rates are evaluated in the subjects with naïve, those with once treatment failure experience, those with twice treatment failure experience, those with thrice treatment failure experience, those with four-time treatment failure experience, and those with five-time treatment failure experience, respectively. The investigators define successful eradication as a negative 13C-urea breath test at least four weeks after the completion of H. pylori eradication and discontinuation of antibiotics and proton pump inhibitors. The eradication rates are determined by ITT and PP analyses. The ITT analysis evaluates all enrolled participants. The PP analysis evaluates those who take >= 80% of the study medications and receive post-treatment 13C-urea breath test. The staffs assessing antibiotic sensitivity and the 13C-urea breath test are blinded.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chi Cheng, MD, PhD, Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischbach L, Evans EL. Meta-analysis: the effect of antibiotic resistance status on the efficacy of triple and quadruple first-line therapies for Helicobacter pylori. Aliment Pharmacol Ther. 2007 Aug 1;26(3):343-57. doi: 10.1111/j.1365-2036.2007.03386.x. PMID 17635369